CLINICAL TRIAL: NCT01046201
Title: Pediatric Obesity Research Registry
Acronym: PORR
Status: Withdrawn | Type: Observational
Why Stopped: To revise protocol for a more concise inclusion/exclusion criteria
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Don P. Wilson, MD, Phoenix Children's Hospital
Other Study IDs: 09-034
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2011-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese Children

SUMMARY:
The Pediatric Obesity Research Registry will function to collect and catalog historical and medical chart related clinical data of patients presenting with pediatric obesity and who agree to participate.

DETAILED DESCRIPTION:
Individuals between age 1 and 18 years who present to the endocrinology clinic for management of elevated BMI/Obesity (Body Mass Index≥95th percentile of age and gender), will be given the opportunity to read the consent form, have any questions/ concerns addressed prior to obtaining informed consent from the research team (consisting of the PI and the Co-investigators) who are also part of the child's clinical care team. The child's clinician will introduce the study to the parents. The Investigator will obtain written informed consent from the child's parents. The clinical care team/research registry investigators will address any questions and concerns prior to obtaining written informed consent and any future questions and concerns. In this manner, Patients seen at the Phoenix Children's Hospital (PCH) Division of Endocrinology and Diabetes with an obesity diagnosis will be asked to provide their written informed consent to allow their past, current and future identifiable medical record information related to their obese condition to be placed in the Pediatric Obesity Research Registry.

For individuals who respond to Potential advertisement or who contact the research team over the phone, a verbal explanation will be given over the phone and an offer to send a copy of the consent via mail/fax/email, and if interested scheduling a follow up appointment. At the clinic visit, the above noted procedure will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between age 1 and 18 years who present to the endocrinology clinic for management of elevated BMI/Obesity
* Individuals between age 1 and 18 years who respond to advertisement or who contact the research team over the phone, for management of elevated BMI/Obesity (Body Mass Index ≥ 95th percentile of age and gender)

Exclusion Criteria:

* A Body Mass Index less than 95th percentile of age and gender

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Obese patients up to age 18 years treated at Phoenix Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donnie P. Wilson, MD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States